CLINICAL TRIAL: NCT06992986
Title: Urinary Microbiome Differences in Bladder Cancer, Benign Urinary Diseases and Healthy Counterpars Adult Male Population: a Pilot Study
Brief Title: Urinary Microbiome Differences in Bladder Cancer, Benign Urinary Diseases and Healthy Counterparts in Adult Male Population
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS91/IRE/24
Record Dates: First submitted 2025-03-18; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples and tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with malignant disease: Will include 30 patients with tumor pathology (10 non-muscle-invasive and 20 muscle-invasive) in which urine samples will be analyzed and, tissue from radical cystectomy samples, will be used to evaluate the urinary microbiome.
  Interventions: Other: Investigating differences in the bladder microbiome
- Non-pathological control subjects/"healthy" controls: Healthy controls will be selected from men with an age within the above-mentioned range, not affected by urinary pathology and/or other overt pathology.
  Suitable controls will be recruited from the institution's staff and/or visiting for occupational medicine.
  Interventions: Other: Investigating differences in the bladder microbiome
- Control patients with "benign" pathologies: This cohort will include individuals with renal cysts, benign prostatic obstruction, ureteropyelic or ureteral obstruction, undergoing surgical therapy.
  The same exclusion criteria as cohort 2 apply.
  Interventions: Other: Investigating differences in the bladder microbiome

INTERVENTIONS:
Other: Investigating differences in the bladder microbiome — Urine samples and tissue from radical cystectomy specimens will be analyzed for the assessment of the urinary microbiome.
  The 16s rRNA gene will be amplified and the resulting amplicons analyzed by Illumina sequencing. To distinguish contaminants, DNA from the sample will be quantified by qPCR and compared to a known urine sample of E. coli. DNA will be extracted using the Quiagen kit and stored at -20 °C until PCR amplification. Bacterial DNA will be amplified with specific primers covering the V1-V3 hypervariable region of the 16S rRNA gene. Libraries will be prepared using the Illumina 16S microbiome sequencing protocol, and their quality will be verified by Bioanalyzer and quantity by qPCR. Sequencing will be performed in "paired-end" mode on Illumina sequencers. Alpha, beta diversity and species richness will be measured.

SUMMARY:
The study aims to investigate alterations in the bladder microbiome in adult men with bladder cancer, healthy men, and men with benign urinary disease

DETAILED DESCRIPTION:
The presence of diverse bacterial representations characterizes a healthy microbiome in both men and women. Differences in bacterial diversity and richness have been observed in subjects with bladder cancer. Investigating the complex relationship between the urinary microbiome and bladder cancer is imperative and requires extensive exploration. The urinary microbiome in patients with bladder cancer has shown high variability in results between studies.

These differences may suggest an interaction with bladder tissue and a potential association; however, it is still unclear whether this association precedes or follows bladder cancer. Regarding phylum-level representations, an abundance of Proteobacteria and Corynebacterium, and a decreased abundance of the genera Ruminococcus and Bifidobacterium have been identified in patients with bladder cancer. The latter two are considered anti-inflammatory bacteria important for mucosal homeostasis. Furthermore, with regard to tumor grade, an increase in Veillonella has been reported in pTa/T1Hg, CIS and T2 tumors; Corynebacterium and Staphylococcus are increased in high-grade NMIBC and low-grade pTa tumors, respectively.

The study aims to investigate possible differences in bacterial representations in patients with bladder cancer, patients with benign urinary diseases and healthy subjects.

Furthermore, possible variations in bacterial profiles in patients with bladder cancer based on tumor stage will be investigated.

differences in bacterial representations in patients with bladder cancer, patients with benign urinary diseases and healthy subjects. In addition to possible variations in bacterial profiles in patients with bladder cancer based on tumor stage.

ELIGIBILITY:
Inclusion Criteria (Bladder Cancer Patients):

* Diagnosis of bladder cancer
* Negative urine culture
* Histological confirmation of urothelial carcinoma
* Patients undergoing radical cystectomy

Exclusion Criteria:

* Presence of other neoplasias
* History of previous BCG therapy
* Use of indwelling catheter
* Active antibiotic treatment with two months prior to participation
* History of sexual transmitted diseases
* Presence of chronic intestinal inflammation
* Previous neoadyuvant therapy

Inclusion Criteria Controls No-Pathologic/Healthy):

- Controls will be collected from men within the specified age range. Eligible controls may be drawn from the institution's personnel attending the occupational medicine department or in service in the Institute.

Exclusion Criteria:

* Diabetes
* Chronic Kidney Disease
* Cardiac disease
* Hepatic disease

Inclusion Criteria(Benign Urinary Disease)

-To ensure that alterations in the microbiome observed in bladder cancer patients are unique to this condition, an additional group with benign urinary diseases will be included in the analysis. This group will encompass individuals with renal cysts, benign prostatic obstruction, ureteropelvic or ureteral obstruction undergoing surgical therapy.

Exclusion Criteria:

* NA

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by bladder cancer, no pathologic/healthy and patients with benign urinary disease.
  * Men
  * Fifty to seventy years of age
  * Written informed consent provided
  * compliants subjects able to follow the study protocol
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-07-06 (Estimated); Study Completion 2025-07-06 (Estimated)

PRIMARY OUTCOMES:
Differences in the bladder microbiome | 36 months
  To investigate differences in the bladder microbiome in men with bladder cancer, healthy men, and men with benign urinary disease. The study involves collecting urine using a mid-stream clean-catch technique.
  Subsequent DNA extraction, sequencing, and identification will allow the study of the bacteria within the samples. In this way, variations in bacterial profiles between patients will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Simone, Doctor, Principal Investigator — IRCCS National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided